CLINICAL TRIAL: NCT06633133
Title: Comparing the Safety and Efficacy of Virtual Ileostomy Versus Diverting Ileostomy in Patients Undergoing Total Mesorectal Excision for Rectal Cancer: a Multicentre, Prospective, Open-label, Blinded Endpoint, PROBE Study
Brief Title: Virtual Ileostomy Versus Diverting Ileostomy in Patients Undergoing Total Mesorectal Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VIRTUAL 01
Record Dates: First submitted 2024-09-29; First posted 2024-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: virtual ileostomy; diverting ileostomy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual ileostomy (Experimental): A pre-stage ileostomy, anchored under the abdominal wall by a vascular sling or rubber tape through the mesenteric window, is delivered to the outside of the abdomen, where the VI is pulled through the abdominal wall.
  Interventions: Procedure: Virtual ileostomy
- Diverting ileostomy (No Intervention): Diverting ileostomy (DI) is a common fecal diversion procedure performed in patients undergoing total mesorectal excision (TME) procedure for rectal cancer to protect the anastomosis and reduce the risk of complications.

INTERVENTIONS:
Procedure: Virtual ileostomy — A pre-stage ileostomy, anchored under the abdominal wall by a vascular sling or rubber tape through the mesenteric window, is delivered to the outside of the abdomen, where the VI is pulled through the abdominal wall.
  Arms: Virtual ileostomy

SUMMARY:
The goal of this clinical trial is to learn to compare the safety and efficacy of virtual ileostomy versus diverting ileostomy in patients undergoing sphincter-saving surgery for rectal cancer. The main questions it aims to answer are:

* Is the virtual ileostomy a safe and effective alternative to the ileostomy?
* Is it scientifically reasonable to perform diverting ileostomy intraoperatively? Researchers will compare virtual ileostomy to diverting ileostomy to see if the virtual ileostomy works to reduce rates of stoma.

Participants will:

* Performing diverting ileostomy or virtual ileostomy undergoing sphincter-saving surgery for rectal cancer
* Continuous follow-up of their complications after the first surgery

DETAILED DESCRIPTION:
This study is a national multicenter, large-sample, randomized controlled study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rectal cancer confirmed by pathology
* Age ≥ 18 years
* Total mesorectal excision (TME) surgical procedures and colon-rectum or colon-anal anastomosis：1.anterior resection (AR/ PME), 2. low anterior resection (LAR) , 3.intersphincteric abdominoperineal resection (ISR), 4.transanal total mesorectal excision (TaTME)
* Signed informed consent
* Ability to understand the nature and risks of participating in the trial

Exclusion Criteria:

* Emergency surgery, open surgery
* ASA score >3points
* Patients with combined complete intestinal obstruction
* Long-term history of using immunosuppressants or glucocorticoids
* Combined severe cardiac disease: with congestive heart failure or NYHA cardiac function ≥ grade 2. Patients with a history of myocardial infarction or coronary artery surgery within 6 months before the procedure
* Chronic renal failure (requiring dialysis or glomerular filtration rate <30 mL/min)
* Intraoperative combined multi-organ resection
* Combined cirrhosis of the liver
* Intraoperative findings of incomplete anastomosis and positive insufflation test
* Modified Bacon procedure(Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis)
* Due to an intraoperative accident the surgeon felt that a diverting ileostomy was necessary.
* Currently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication index (CCI) at the 6th postoperative month | An average of 6 month from the date of low anterior resection for rectal cancer until the date of when the patient's condition is stabilized without complications
  The Comprehensive Complication Index (CCI)summarises all postoperative complications based on the established Clavien-Dindo classification (ranging from mild complications not leading to a deviation from the normal clinical course (grade I) up to postoperative death (grade V)) at an individual patient level according to their grade of severity.

SECONDARY OUTCOMES:
Comprehensive Complication Index (CCI) at the first postoperative, 3 months postoperative, 1 year postoperative,3 years postoperative,5 years postoperative | 5 year
  The Comprehensive Complication Index (CCI)summarises all postoperative complications based on the established Clavien-Dindo classification (ranging from mild complications not leading to a deviation from the normal clinical course (grade I) up to postoperative death (grade V)) at an individual patient level according to their grade of severity.
First postoperative complications | From the date of randomization until the date of discharge, an average of 7 to 14 days
  First postoperative complications(including abdominal abscess, peritonitis, anastomotic leakage, anastomotic bleeding, pelvic infection, surgical incision infection, peritonitis, anastomotic stenosis, intestinal obstruction, peri-wound complications, incisional hernia, and others) based on the established Clavien-Dindo classification (ranging from mild complications not leading to a deviation from the normal clinical course (grade I) up to postoperative death (grade V)) at an individual patient level according to their grade of severity.
Stoma-related complications | Through study completion, an average of 5 year
  Wounds/abscesses/edema/dermatitis/ulcers around the diverting Ileostomy; parastomal hernia; stoma prolapse; acute kidney injury; dehydration/output >1500 mL/day； other stoma-related complications
Complications after ileostomy closure | Through study completion, an average of 5 year
  Anastomotic leakage； intestinal anastomotic leakage； anastomotic stenosis; bowel obstruction; other wound complications （Wound dehiscence/bleeding/sinus tract/abscess/fat liquefaction）; burst abdomen (dehiscence of abdominal fascia); incisional hernia; fecal incontinence; reoperation; other complications
Postoperative hospitalization days(Initial and all subsequent hospitalizations) | Through study completion, an average of 5 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded days of postoperative hospitalization after low anterior resection for rectal cancer, if the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record days of postoperative hospitalization due to complications and/or reoperation since the data of low anterior resection for rectal cancer.
The number of hospitalizations(Initial and all subsequent hospitalizations) | Through study completion, an average of 5 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded the number of hospitalizations after low anterior resection for rectal cancer. If the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the number of hospitalization due to complications and/or reoperation since the data of low anterior resection for rectal cancer.
Duration of bearing the stoma (months) | Through study completion, an average of 5 year
  If the virtual stoma group required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the duration of bearing the stoma since the data of surgery of diverting ileostomy.
Total hospitalization costs(Initial and all subsequent hospitalizations) | Through study completion, an average of 5 year
  Patients in the virtual stoma group who did not have a second surgery due to complications recorded the costs after the first surgery for rectal cancer, if the virtual stoma group required bedside or secondary surgery for converted to diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the costs due to complications and reoperation since the data of the first surgery for rectal cancer.
Number of participants with terminal ostomy | Through study completion, an average of 5 year
  Hartmann's procedure or for example, abdominoperineal extirpation，and transverse colostomy
Number of Participants with unscheduled secondary surgery | Through study completion, an average of 5 year
  Patients performed unscheduled secondary surgery due to complications.
The rate at which virtual ileostomy was converted to diverting ileostomy | Through study completion, an average of 5 year
  The virtual ileostomy group required bedside or secondary surgery to convert to diverting ileostomy due to complications
Virtual ileostomy remove time(days) | During hospitalization,approximately 14 days
  Duration of days from the date of radical resection of rectal cancer to virtual stoma removed.
Bile acid concentration of drainage fluid | During hospitalization,approximately 7 days
  The investigators are monitoring the concentration of bile acids in the first postoperative drainage fluid.
Number of participants with stoma (terminal/loop) at 6 months after initial surgery | 6 months from the date of first surgery for rectal cancer
  Patients carrying stoma 6 months after the first surgery for rectal cancer
Interventional drainage rate | Through study completion, an average of 5 year
  Patient requires interventional drainage due to complications.
Fecal Incontinence Scale(Wexner Score) | Through study completion, an average of 5 year
  The defecation function of all postoperative patients. Wexner score range is 0-20 points, with 0 points indicating normal and 20 points indicating complete incontinence.
Quality of life(EORTC QLQ-C30) | Through study completion, an average of 5 year
  The quality of life of all patients was assessed using relevant scales[EORTC (The European Organization for Reasearch and Treatment of Cancer) QLQ-C30(Quality of Life Questionnare-Core 30)]. The EORTC QLQ-C30 (V3. O) consists of 30 entries, which can be divided into 15 domains, including 5 functional domains (physical, role, cognitive, emotional, and social functions), 3 symptom domains (fatigue, pain, nausea, and vomiting), 1 overall health/quality of life domain, and 6 individual entries (each as a domain). EORTC QLQ-C30 has a total of 30 entries. Among them, entries 29 and 30 are divided into seven levels, ranging from 1 to 7 points based on their answer options; the other entries are divided into 4 levels: none(1 point), a little（2 points）, more（3 points）, many（4 points）. The QLQ-C30 scale is reversed except for items 29 and 30 (the higher the value, the worse the quality of life).
Disease free survival (DFS) | Through study completion, an average of 5 year
  Disease free survival
Overall survival (OS) | Through study completion, an average of 5 year
  Overall survival
Rate of permanent ileostomy | From the date of first surgery,an average of 3 year
  Patients who underwent diverting Ileostomy were converted to permanent ileostomy.
Completion of intended perioperative or adjuvant chemotherapy | Through study completion, an average of 5 year
  Completion of intended perioperative or adjuvant chemotherapy
Low anterior resection syndrome for rectal cancer | Through study completion, an average of 5 year
  The investigators use LARS scale to evaluate the patient's defecation function.The LARS rating scale consists of 5 questions: voiding incontinence, fluid voiding incontinence, frequency of voiding, voiding aggregation, and voiding urgency. 0-20 is classified as no LARS, 21-29 is classified as mild LARS, 30-42 is classified as severe LARS.
Quality of life for fecal incontinence | Through study completion, an average of 5 year
  The Fecal Incontinence Quality of Life Scale (FIQL) is mainly used to evaluate the quality of life of patients with fecal incontinence. It includes four main aspects: lifestyle changes, psychological coping/behavioral limitations, depression/self-perception, and social embarrassment. The FIQL is analyzed as a total score; the higher the patient's score, the higher the patient's quality of life.
Permanent ileostomy rate | 3 years from the date of first surgery for rectal cancer
  Patients with diverting ileostomy who underwent sphincter-saving surgery for rectal cancer were converted to permanent ileostomy.
Mortality | 30 days from the date of first surgery for rectal cancer
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: fan li, Study Chair — Daping Hospital, Third Military Medical University
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degiuli M, Elmore U, De Luca R, De Nardi P, Tomatis M, Biondi A, Persiani R, Solaini L, Rizzo G, Soriero D, Cianflocca D, Milone M, Turri G, Rega D, Delrio P, Pedrazzani C, De Palma GD, Borghi F, Scabini S, Coco C, Cavaliere D, Simone M, Rosati R, Reddavid R; collaborators from the Italian Society of Surgical Oncology Colorectal Cancer Network Collaborative Group. Risk factors for anastomotic leakage after anterior resection for rectal cancer (RALAR study): A nationwide retrospective study of the Italian Society of Surgical Oncology Colorectal Cancer Network Collaborative Group. Colorectal Dis. 2022 Mar;24(3):264-276. doi: 10.1111/codi.15997. Epub 2021 Dec 6. PMID 34816571
- [Background] Zhao S, Zhang L, Gao F, Wu M, Zheng J, Bai L, Li F, Liu B, Pan Z, Liu J, Du K, Zhou X, Li C, Zhang A, Pu Z, Li Y, Feng B, Tong W. Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Laparoscopic Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1151-1158. doi: 10.1001/jamasurg.2021.4568. PMID 34613330
- [Background] Lightner AL, Vogel JD, Carmichael JC, Keller DS, Shah SA, Mahadevan U, Kane SV, Paquette IM, Steele SR, Feingold DL. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Surgical Management of Crohn's Disease. Dis Colon Rectum. 2020 Aug;63(8):1028-1052. doi: 10.1097/DCR.0000000000001716. No abstract available. PMID 32692069
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; TaTME Registry Collaborative. Transanal Total Mesorectal Excision: International Registry Results of the First 720 Cases. Ann Surg. 2017 Jul;266(1):111-117. doi: 10.1097/SLA.0000000000001948. PMID 27735827
- [Background] Palumbo P, Usai S, Pansa A, Lucchese S, Caronna R, Bona S. Anastomotic Leakage in Rectal Surgery: Role of the Ghost Ileostomy. Anticancer Res. 2019 Jun;39(6):2975-2983. doi: 10.21873/anticanres.13429. PMID 31177138
- [Background] Huttner FJ, Probst P, Mihaljevic A, Contin P, Dorr-Harim C, Ulrich A, Schneider M, Buchler MW, Diener MK, Knebel P. Ghost ileostomy versus conventional loop ileostomy in patients undergoing low anterior resection for rectal cancer (DRKS00013997): protocol for a randomised controlled trial. BMJ Open. 2020 Oct 15;10(10):e038930. doi: 10.1136/bmjopen-2020-038930. PMID 33060088
- [Background] Sacchi M, Legge PD, Picozzi P, Papa F, Giovanni CL, Greco L. Virtual ileostomy following TME and primary sphincter-saving reconstruction for rectal cancer. Hepatogastroenterology. 2007 Sep;54(78):1676-8. PMID 18019692
- [Background] Baloyiannis I, Perivoliotis K, Diamantis A, Tzovaras G. Virtual ileostomy in elective colorectal surgery: a systematic review of the literature. Tech Coloproctol. 2020 Jan;24(1):23-31. doi: 10.1007/s10151-019-02127-2. Epub 2019 Dec 9. PMID 31820192
- [Background] Zenger S, Gurbuz B, Can U, Balik E, Yalti T, Bugra D. Comparative study between ghost ileostomy and defunctioning ileostomy in terms of morbidity and cost-effectiveness in low anterior resection for rectal cancer. Langenbecks Arch Surg. 2021 Mar;406(2):339-347. doi: 10.1007/s00423-021-02089-w. Epub 2021 Feb 4. PMID 33537875
- [Background] Miccini M, Amore Bonapasta S, Gregori M, Barillari P, Tocchi A. Ghost ileostomy: real and potential advantages. Am J Surg. 2010 Oct;200(4):e55-7. doi: 10.1016/j.amjsurg.2009.12.017. PMID 20887836
- [Background] Cerroni M, Cirocchi R, Morelli U, Trastulli S, Desiderio J, Mezzacapo M, Listorti C, Esperti L, Milani D, Avenia N, Gulla N, Noya G, Boselli C. Ghost Ileostomy with or without abdominal parietal split. World J Surg Oncol. 2011 Aug 18;9:92. doi: 10.1186/1477-7819-9-92. PMID 21849090
- [Background] Mori L, Vita M, Razzetta F, Meinero P, D'Ambrosio G. Ghost ileostomy in anterior resection for rectal carcinoma: is it worthwhile? Dis Colon Rectum. 2013 Jan;56(1):29-34. doi: 10.1097/DCR.0b013e3182716ca1. PMID 23222277
- [Background] McKechnie T, Lee J, Lee Y, Tessier L, Amin N, Doumouras A, Hong D, Eskicioglu C. Ghost Ileostomy Versus Loop Ileostomy Following Oncologic Resection for Rectal Cancer: A Systematic Review and Meta-Analysis. Surg Innov. 2023 Aug;30(4):501-516. doi: 10.1177/15533506231169066. Epub 2023 Apr 4. PMID 37013791
- [Background] Flor-Lorente B, Sanchez-Guillen L, Pellino G, Frasson M, Garcia-Granero A, Ponce M, Domingo S, Paya V, Garcia-Granero E. "Virtual ileostomy" combined with early endoscopy to avoid a diversion ileostomy in low or ultralow colorectal anastomoses. A preliminary report. Langenbecks Arch Surg. 2019 May;404(3):375-383. doi: 10.1007/s00423-019-01776-z. Epub 2019 Mar 27. PMID 30919049